CLINICAL TRIAL: NCT01714999
Title: A Prospective Evaluation of the Current Treatment Regime for Acute Traumatic Laceration of the Olecranon and Prepatellar Bursa
Brief Title: Treatment of Acute Traumatic Laceration of the Olecranon and Prepatellar Bursa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sebastian. F. Baumbach, M.D., Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 415-12; 1692/2012 (Other: Ethics commission Medical University of Vienna)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Traumatic Laceration of the Olecranon or Prepatellar Bursa
Keywords: olecranon; prepatellar; bursa; trauma; laceration; bursectomy; bursa reconstruction
MeSH Terms: conditions — Wounds and Injuries; Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bursectomy: Vienna (Experimental): At the Department of Trauma Surgery, Medical University of Vienna, bursectomy is considered the gold standard in case of traumatic laceration of the OB or PB bursa.
  Interventions: Procedure: Bursectomy
- Bursal reconstruction: Munich (Experimental): At the Department of Trauma Surgery, Medical University of Munich, the treatment regime is a primary bursa-preserving therapy.
  Interventions: Procedure: Bursal reconstruction

INTERVENTIONS:
Procedure: Bursectomy — Bursectomy of the OB and PB are performed in the operation theatre under sterile conditions. In case of a laceration of the OB a leash, in case of PB a redon drainage (Charr. 10) is inserted. After application of a sterile bandage a cast is applied in both cases. Patient will receive AB for 5 days, the affected limb will be immobilized until removal of the stiches after 12-14 days.
  Other Names: Removal of the Bursa, Excision of the Bursa
  Arms: Bursectomy: Vienna
Procedure: Bursal reconstruction — The bursal laceration is treated within in ER setting. The wound is cleaned and thoroughly washed, if needed the wound margins are excised. The wound is then closed using simple suture and a plaster applied and removed 5 days later. Antibiotics are be administered for 5 days
  Other Names: Reconstruction of the bursa
  Arms: Bursal reconstruction: Munich

SUMMARY:
Following a recent publication by the authors [1], there is no standardized treatment regime for the treatment of lacerations of the olecranon or prepatellar bursa, although primary bursectomy seems to be the most common treatment regime in Germany, Austria and Switzerland. The aim of this study is to prospectively follow patients who suffered from an acute traumatic laceration of the OB or PB treated, according to the local standards, either by bursectomy (Vie, AT) or bursal reconstruction and direct wound closure (Muc, GER).

[1] Baumbach et al. Evaluation of the current treatment concepts in Germany, Austria and Switzerland for acute traumatic lesions to the prepatellar and olecranon bursa. Injury (2012)

DETAILED DESCRIPTION:
A fall onto the elbow or knee often results in a laceration of the olecranon (OB) and prepatellar bursa (PB), due to their exposed and superficial location. Although a common injury, the authors are not aware of any study dealing with this entity. In order to get a first idea on the treatment concepts currently used, the authors conducted a international online survey among orthopaedic and trauma surgeons in Germany, Austria and Switzerland [1]. The primary treatment approach of more than 70% of Austrian and German surgeons was bursectomy and immobilization, which was performed by less than 50% of Swiss physicians.

At the Departments of Trauma Surgery of the Medical University of Vienna and of the Medical University of Munich, two opposing treatment concepts are being practised. Whereas in Vienna a bursectomy is performed in case of traumatic laceration of the OB and PB, a primary bursal reconstruction is performed at the Medical University of Munich.

The aim of this study is to prospectively follow patients who suffered from an acute traumatic laceration of the OB or PB treated, according to the local standards, either by bursectomy (Vie, AT) or bursal reconstruction and direct wound closure (Muc, GER).

The Hypothesis of this study is, that there is no difference with respect to complications between bursectomy and bursal reconstruction in case of acute traumatic laceration of the OB and PB.

1. Baumbach et al. Evaluation of the current treatment concepts in Germany, Austria and Switzerland for acute traumatic lesions to the prepatellar and olecranon bursa. Injury (2012)

ELIGIBILITY:
Inclusion Criteria:

* Acute lacerations of the OB or PB (<12h)
* Age 18 - 60 years
* Patient can read and understand German

Exclusion Criteria:

* Immunodeficient patients
* Severe dementia
* Chronic alcoholism
* Conditions affecting the neuromuscular- or musculoskeletal system
* Previous surgical interventions at the same joint
* Conditions affecting wound healing (including chronic alcoholism, insulin dependent diabetes
* Neurological diseases
* Patient is not available for follow-up visits
* Patient suspected to be non-compliant
* No major concomitant injuries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Wound infection | 6 weeks

SECONDARY OUTCOMES:
Bursitis | 12 month

OTHER OUTCOMES:
Treatment costs of a standard patient | 6 weeks / 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian F Baumbach, MD, Principal Investigator — Ludwig-Maximilians - University of Munich; Vikoria Bogner, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (2):
- Department of Trauma Surgery, Medical University of Vienna, Vienna, Austria
- Department of Trauma Surgery, Medical University of Munich, Munich, Germany

REFERENCES:
- [Background] Baumbach SF, Domaszewski F, Wyen H, Kalcher K, Mutschler W, Kanz KG. Evaluation of the current treatment concepts in Germany, Austria and Switzerland for acute traumatic lesions to the prepatellar and olecranon bursa. Injury. 2013 Nov;44(11):1423-7. doi: 10.1016/j.injury.2012.08.008. Epub 2012 Sep 11. PMID 22980398